CLINICAL TRIAL: NCT01642134
Title: PHASE IV Study of Dual Antiplatelet Therapy Versus Oral Anticoagulation for a Short Time to Prevent Cerebral Embolism After Percutaneous Aortic Valve Implantation. Multicenter Randomized Clinical Trial
Brief Title: Dual Antiplatelet Therapy Versus Oral Anticoagulation for a Short Time to Prevent Cerebral Embolism After TAVI
Acronym: AUREA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Andres Iñiguez Romo, MD, PhD (Other Government)
Responsible Party: Sponsor-Investigator, Andres Iñiguez Romo, MD, PhD, MD; PHD, Hospital de Meixoeiro
Organization: Hospital de Meixoeiro (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEIX-VALV-001; 2011-005784-24 (EudraCT Number)
Record Dates: First submitted 2012-06-19; First posted 2012-07-17 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Aortic Valve Stenosis; Stroke
Keywords: Antiplatelet; Anticoagulation
MeSH Terms: conditions — Aortic Valve Stenosis; Stroke | interventions — Aspirin; Clopidogrel; Acenocoumarol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duoplavin (Active Comparator): Both active substances in DuoPlavin: clopidogrel and acetylsalicylic acid, are inhibitors of platelet aggregation. Clopidogrel stops the platelets aggregating by blocking ADP. Acetylsalicylic acid the platelets aggregating by blocking the prostaglandin cyclo oxygenase.
  Interventions: Drug: aspirin+clopidogrel (Duoplavin)
- acenocumarol (Sham Comparator)
  Interventions: Drug: aspirin+clopidogrel (Duoplavin)

INTERVENTIONS:
Drug: aspirin+clopidogrel (Duoplavin) — 100 mg aspirin ;75 mg clopidogrel 3º months
  Other Names: DUOPLAVIN (aspirin 100 mg + clopidogrel 75 mg).; SINTROM (ACENOCUMAROL).

SUMMARY:
The purpose of this study is to determine the incidence of major vascular events (ischemic or haemorrhagics) at the third month after initiation of the antithrombotic treatment (oral anticoagulation or dual antiplatelet therapy) in both arms followed TAVI.

DETAILED DESCRIPTION:
Transcatheter aortic valve implantation (TAVI) procedure using any of their vascular access is an option with proven benefit definitively for treatment of severe symptomatic aortic stenosis in patients considered unsuitable for conventional open heart surgery.

By avoiding the hemodynamic effects, cardiovascular and cerebral microembolic load of cardiopulmonary bypass circulation, it is assumed that the TAVI procedure is beneficial despite the risk of neurological complications. Currently antithrombotic therapy after the procedure is not standardized. International treatment guidelines recommends that post-operative patients with a conventional surgical aortic bioprosthesis maintain oral anticoagulation for 3 months after the procedure, unless otherwise noted for its continuation. Whereas some studies have postulated that in patients with aortic bioprostheses, dual antiplatelet therapy is as effective to prevent major cardiac and cerebrovascular events as oral anticoagulation, with a lower incidence of bleeding complications at 3 months of treatment, the investigators formulated the following hypothesis:

• There is a lower incidence of major cardiac and cerebrovascular events in patients with dual antiplatelet therapy compared to patients with oral anticoagulation for 3 months after implantation of an aortic bioprosthesis TAVI procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (more than 18 years) with ability to understand and accept the participation in the clinical trial.
2. Patients with symptomatic degenerative severe aortic stenosis rejected for conventional surgical aortic valve replacement due to unacceptably high risk and accepted for TAVI procedure
3. Signed informed consent.
4. Patients who are not participating in any other clinical trial or research study.

Exclusion Criteria:

1. Patients under oral anticoagulation treatment
2. Patients who can not undergo MRI study
3. Recent stroke < 14 days prior, revascularized coronary artery disease or life expectancy < 12 months
4. Patients with proven allergy to aspirin, clopidogrel or acenocoumarol
5. Patients that after TAVI procedure can not undergo a regimen of dual antiplatelet therapy or oral anticoagulation for 3 months due to any new post-TAVI medical indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-04; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of dual antiplatelet therapy versus oral anticoagulation for prevention of cerebral thromboembolism by the detection of new areas of cerebral infarction by Magnetic Resonance Imaging (MRI) 3 months after TAVI. | 3 months

SECONDARY OUTCOMES:
Determine the incidence of new areas of cerebral infarction by MRI between the different routes of vascular access and the various valve devices. | 1 hour before TAVI, 1 hour and 24 hours after TAVI
Identify the development of cognitive impairment after TAVI | Pre-TAVI, and at 1º 3º and 6º month after TAVI
  By the application of: 1)Mini-Mental State Examination (MMSE); 2)SF 36 (spanish version); 3)The NIHSS (National Institute of Health Stroke Scale). The evaluation of the neurological tests will be performed by a certificated neurologist.
Evaluate the Quality of life after TAVI. | Pre-TAVI, and at 1º; 3º and 6º month after TAVI.
  By the application of Euroquol EQ5.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Iniguez Romo, MD;PHD, Principal Investigator — Hospital Universitario Alvaro Cunqueiro; Victor A. Jimenez Diaz, MD;Msc, Principal Investigator — Hospital clinico universitario Vigo; Mariano Larman Tellechea, MD, Principal Investigator — Policlínica de Guipuzcoa SA San Sebastián; Pablo Juan Salvadores, Pharma,MPH, Study Director — Hospital Universitario Álvaro Cunqueiro; Jose M. Hernandez, MD, Principal Investigator — Hospital Virgen de la Victoria
Locations (4):
- Spain (4):
  - Policlínica de Guipuzcoa.SA, San Sebastián, Guipúzcoa
  - Hospital Universitario Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital clinico Universitario Bellvitge, Barcelona
  - Hospital Clinico Universitario de Malaga, Málaga

REFERENCES:
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Kahlert P, Knipp SC, Schlamann M, Thielmann M, Al-Rashid F, Weber M, Johansson U, Wendt D, Jakob HG, Forsting M, Sack S, Erbel R, Eggebrecht H. Silent and apparent cerebral ischemia after percutaneous transfemoral aortic valve implantation: a diffusion-weighted magnetic resonance imaging study. Circulation. 2010 Feb 23;121(7):870-8. doi: 10.1161/CIRCULATIONAHA.109.855866. PMID 20177005
- [Background] Herrmann M, Vos P, Wunderlich MT, de Bruijn CH, Lamers KJ. Release of glial tissue-specific proteins after acute stroke: A comparative analysis of serum concentrations of protein S-100B and glial fibrillary acidic protein. Stroke. 2000 Nov;31(11):2670-7. doi: 10.1161/01.str.31.11.2670. PMID 11062293
- [Background] Dunning J, Versteegh M, Fabbri A, Pavie A, Kolh P, Lockowandt U, Nashef SA; EACTS Audit and Guidelines Committee. Guideline on antiplatelet and anticoagulation management in cardiac surgery. Eur J Cardiothorac Surg. 2008 Jul;34(1):73-92. doi: 10.1016/j.ejcts.2008.02.024. Epub 2008 Mar 28. PMID 18375137
- See also: Related Info — http://www.cardiologia-vigo.com/